CLINICAL TRIAL: NCT01204801
Title: Randomized Pivotal Trial to Assess the Safety and Efficacy of Preoperative Focused Microwave Thermotherapy Plus Preoperative Chemotherapy Versus Preoperative Chemotherapy Alone for Cytoreduction of Large Breast Cancer in Female Patients With Intact Breast
Brief Title: Randomized Study of Combination Chemotherapy With or Without Focused Microwave Thermotherapy Before Surgery in Treating Women With Large Breast Cancer Tumors
Acronym: Medifocus301
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medifocus, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102-00-301
Record Dates: First submitted 2010-08-26; First posted 2010-09-17 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Cancer; Breast Cancer; Breast Tumor; Breast Neoplasm; Neoplasms by Site; Neoplasms; Breast Diseases; Breast Conserving Surgery; Breast Conservation; Partial Mastectomy; Lumpectomy; Mastectomy; Surgery; Neoadjuvant Therapy; Primary Therapy; Neoadjuvant Systemic Therapy; Thermotherapy; Fever Therapy; Hot Temperature; Hyperthermia; Hyperthermia, Therapeutic; Hyperthermia, Local; Hyperthermia, Induced; Therapeutic Hyperthermia; Microwave; Focused Microwave; Focused Microwave Thermotherapy; Minimally Invasive; Doxorubicin; Epirubicin; Epidoxirubicin; Immunosuppresive Agent; Immunologic Factors; Physiological Effects of Drugs; Chemotherapy; Drug Therapy; Pharmalogic Actions; Antirheumatic Agents; Therapeutic Uses; Antineoplastic Agents, Alkylating; Alkylating Agents; Molecular Mechanisms of Pharmacological Action; Antineoplastic Agents; Myeloblative Agonists; Antibiotics, Antineoplastic; Anthracycline Agents
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasms by Site; Breast Diseases; Hyperthermia | interventions — Drug Therapy; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thermochemotherapy (Experimental): Preoperative Anthracycline Doxorubicin 60mg/m2 (or Epirubicin 100 mg/m2) + Standard of Care chemotherapy and drugs + Thermotherapy. Thermotherapy at first 3 chemotherapy treatments for Anthracycline chemotherapy nominally every 21±7 days plus Standard of Care chemotherapy.
  Interventions: Device: Focused Microwave Thermotherapy
- Chemotherapy (control) (Active Comparator): Preoperative Anthracycline Doxorubicin 60mg/m2 (or Epirubicin 100 mg/m2) + Standard of Care chemotherapy and drugs
  Interventions: Drug: Chemotherapy (control)

INTERVENTIONS:
Device: Focused Microwave Thermotherapy — Anthracycline Doxorubicin 60mg/m2 (or Epirubicin 100 mg/m2) + Standard of Care chemotherapy and drugs + Thermotherapy. Thermotherapy at first 3 chemotherapy treatments for Anthracycline chemotherapy nominally every 21±7 days plus Standard of Care chemotherapy. (A targeted tumor temperature of 44ºC (plus or minus 1.5ºC) and a targeted thermal dose of 80 equivalent treatment minutes (plus or minus 20 treatment minutes)). In the event that the targeted minimum cumulative thermal dose of 180 equivalent treatment minutes is not achieved in the first three treatments, an optional fourth thermotherapy treatment may be administered in combination with the fourth course of Anthracycline and standard of care chemotherapy. Standard of care (including breast imaging, drugs, and radiation) will be provided to all eligible subjects during and following the above study treatments.
  Other Names: APA-1000 Focused Microwave Thermotherapy Device; Adriamycin
  Arms: Thermochemotherapy
Drug: Chemotherapy (control) — Anthracycline Doxorubicin 60mg/m2 (or Epirubicin 100 mg/m2) + Standard of Care chemotherapy and drugs. Anthracycline chemotherapy nominally every 21±7 days. Standard of care (including breast imaging, drugs, and radiation) will be provided to all eligible subjects during and following the above study treatments.
  Other Names: Adriamycin
  Arms: Chemotherapy (control)

SUMMARY:
The purpose of this randomized Phase III study is to determine whether preoperative focused microwave heat treatment and chemotherapy combined are more effective than preoperative chemotherapy alone in the treatment of large breast cancer tumors in the intact breast. Combining heat with chemotherapy before surgery might shrink the tumor so that it can be removed in a breast conserving surgery (lumpectomy) instead of a mastectomy.

DETAILED DESCRIPTION:
This randomized multicenter Phase III clinical trial is intended to provide histopathological and clinical information on an innovative, minimally-invasive approach (focused microwave thermotherapy) to the preoperative treatment of breast cancer, using a minimally invasive focused microwave phased array device, the Medifocus, Inc. APA 1000 Breast Thermotherapy Treatment System (heat treatment). Subjects with large primary operable breast cancer, in the intact breast, with clinical tumor size greater than or equal to 3.5 cm (including tumor classification T2 or T3), clinically node negative N0 or node positive (N1 or N2) with distant metastasis (M1) or without distant metastasis (M0) will be randomized (ratio 1:1) to receive (1) preoperative thermotherapy combined with preoperative anthracycline-based combination chemotherapy and standard of care versus (2) preoperative anthracycline-based combination chemotherapy and standard of care alone. The anthracycline-based regimen will be limited to those of the current National Comprehensive Cancer Network (NCCN) guidelines for dose/drug/schedule at the time of patient enrollment. In both arms of the study, standard of care including breast imaging, drugs, and radiation therapy will be provided to all eligible subjects during and following the preoperative regimen. At the clinical discretion of the treating physician, subjects that are estrogen-receptor positive may receive Tamoxifen therapy the day following the completion of chemotherapy. Radiation therapy to the breast tissues and lymph nodes will be given as part of the standard of care for eligible subjects. Treatment Arm I (new arm) regimen includes three preoperative thermotherapy treatments at intervals corresponding to the first three cycles of anthracycline-based combination chemotherapy plus standard of care. The addition of preoperative thermotherapy to preoperative anthracycline-based combination chemotherapy may improve the tumor response rate in terms of shrinkage (the primary endpoint) and may increase the option to perform breast conservation (a secondary endpoint) compared to that achieved with preoperative anthracycline-based combination chemotherapy and standard of care alone. Note: Since there is no consensus combination drug regimen for neoadjuvant treatment of large breast cancer tumors, each study site will use its own standard of care which will include other chemotherapy/drug agents commonly used in combination with an anthracycline (Doxorubicin (trade name Adriamycin) or Epirubicin (trade name Ellence)), which is the study base drug type.

The rationale for including patients that have distant metastasis (M1) at enrollment in this study is as follows. Traditionally, patients with stage IV (metastatic) breast cancer and an intact primary breast tumor have been treated with chemotherapy and radiation for palliation of symptoms, because this metastatic condition is considered to be an incurable disease. In some cases, surgery has been considered for stage IV patients with large, symptomatic breast lesions to control local wound complications and to improve quality of life. However, four recent retrospective peer-reviewed studies have suggested that removing the primary tumor may lead to an improvement in overall survival.

The investigator or designee will fully explain the nature of the study to the subject, along with the aims, methods, anticipated benefits, potential hazards and discomfort that participation might entail. After the nature of the study has been explained and all the subject's questions have been answered, and if the subject agrees to participate in the study, the informed consent will be reviewed and signed by the subject.

Each subject will be treated by thermochemotherapy (new arm) or chemotherapy alone (control arm) and followed for 90 days after surgery during the study. Patients will be followed annually as practiced as standard of care by each participating institution - patients will be followed for tumor recurrence and future medical intervention related to the patient's breast cancer.

Thermotherapy is administered in an out-patient setting. During thermotherapy which is completed in approximately 60 minutes or less, the patient is treated in the prone position on a treatment bed. After administering a local anesthetic, to guide the treatment a minimally invasive combination microwave/temperature probe is placed in the tumor under ultrasound guidance. The thermotherapy treatment is adjusted in accordance with patient comfort.

Anthracycline-based chemotherapy will be administered in accordance with standard preoperative chemotherapy delivery at each study center - the number of chemotherapy cycles and cycle timing may vary in this study. Each study center will be using anthracycline (Doxorubicin or Epidoxorubicin) as the base chemotherapy agent and the other chemotherapy agents and drugs will vary depending on the study center and subject specific needs. Each cycle of Doxorubicin at 60 mg/m2 for four cycles or Epidoxorubicin at 100 mg/m2 for 6 cycles and combination Standard of Care chemotherapy will be administered nominally every 21 (plus or minues 7) days. The timing between cycles of anthracycline can be subject specific at the physician's discretion, but in no case will anthracycline be administered with a cycle timing of less than seven (7) days between anthracycline cycles. A thermotherapy session will be administered on the same day as the administration of the first, second, and third cycle of preoperative Doxorubicin or Epidoxorubicin chemotherapy. Chemotherapy will be administered and then the subject will receive thermotherapy. (If the thermotherapy session cannot be administered on the same day as Doxorubicin or Epidoxorubicin chemotherapy it will be administered as soon as possible the following day but no later than 36 hours post Doxorubicin or Epidoxorubicin chemotherapy. The remaining cycle(s) of chemotherapy will then be administered without thermotherapy. If the desired cumulative minimum thermal dose is achieved in the first three thermotherapy treatments, the remaining cycle(s) of chemotherapy will then be administered without thermotherapy. If the desired cumulative minimum thermal dose is not achieved during the first three preoperative Doxorubicin or Epidoxorubicin chemotherapy cycles, thermotherapy will be administered with the fourth cycle of preoperative chemotherapy. If the subject cannot tolerate more than one or two thermotherapy treatments, the subject will continue in the study on the remaining cycles of chemotherapy. If the subject has clinically progressive disease, the thermo-chemotherapy treatment will be discontinued and the subject will receive the remaining cycles of chemotherapy preoperatively or postoperatively (as standard care).

At the end of the course of thermo-chemotherapy or chemotherapy alone, and following all pre-surgery evaluations, the surgeon and subject will make decisions on the extent of surgery to be performed. These decisions will be made on the basis of surgical and institutional standards, and those of the National Comprehensive Cancer Network (NCCN) Breast Cancer Treatment Guidelines. Subjects will undergo mastectomy or breast-conserving surgery. It is understood that some subjects will select mastectomy for treatment even when the surgeon recommends breast conservation. The surgeon shall document the reasons why either mastectomy or breast conservation was selected.

The subject will undergo clinical exam and imaging of the breast to measure tumor size, the day prior to or the day of the lumpectomy or mastectomy. Any additional imaging will be at the discretion of the physician. At the discretion of the physician, an optional core biopsy of the tumor will be taken the day prior or the day of the surgery.

Following surgery, pathology will be performed on the excised breast tumor tissue to determine tumor cell death. For breast conservation, the breast must be of sufficient size to allow adequate tumor removal with a satisfactory cosmetic result. The objective of surgery is to obtain local control of the breast cancer with the best cosmetic result possible. A breast conservation surgery procedure requires excision of the tumor and margins without removal of more normal breast tissue than is required to achieve negative margins. Pathologic evaluation of the excised tissue will determine whether the margins are negative or positive. For subjects with involved margins following breast conservation surgery, if the breast will tolerate it, the subject may undergo one or more further segmental resections in order to achieve clear margins.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must fulfill all of the following criteria to be eligible to participate in the study unless a specific waiver is requested by the investigator, agreed to by the sponsor, and documented for the study records. This protocol does not supersede Institutional IRB requirements for patient eligibility.

  1. Female subject must be 18 years of age or older.
  2. Subject must have adequate cognitive function to understand and sign the IRB/EC - approved informed consent prior to the performance of any study-specific procedure.
  3. The subject must be at no risk for pregnancy either postmenopausal for at least one year, surgically sterile (i.e. hysterectomy), using two forms of birth control one being barrier method or practicing abstinence throughout the length of the study. The subject must also have a negative serum pregnancy test prior to any study-specific procedure.
  4. Subject must have diagnosis by core biopsy of primary breast cancer, invasive ductal carcinoma or invasive lobular carcinoma, clinical tumor size 3.5 cm or greater, tumor classification T2 or T3, clinically node positive (N1, N2) or node negative (N0) by clinical exam, CT scan, or ultrasound, with distant metastasis (M1) or without distant metastasis (M0), with an indication for mastectomy.
  5. Primary tumor must be measurable on breast ultrasound (US).
  6. Primary tumor must be measurable by clinical exam.
  7. Subject is a candidate for mastectomy and is eligible for neoadjuvant treatment.
  8. Subject is a candidate for preoperative anthracycline-based combination chemotherapy.
  9. Subject has a life expectancy of 6 months or more.
  10. Karnofsky Score > 70.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study unless a specific waiver is requested by the investigator, agreed to by the sponsor, and documented appropriately for the study records. This protocol does not supersede Institutional IRB requirements for patient eligibility:

  1. Pregnant or lactating subject.
  2. Mentally unable to participate in the study successfully because they are unable to understand the informed consent or unable to comply with the required study procedures.
  3. Currently has breast implants.
  4. Bilateral breast cancer.
  5. Subjects with malignant breast tumors other than invasive ductal or invasive lobular carcinomas.
  6. Subject is a candidate for breast conservation at enrollment.
  7. Unable to tolerate prone position or breast compression.
  8. Clinically significant heart disease, pacemakers, or defibrillators.
  9. Bleeding disorders. Laboratory evidence of coagulopathy (PT, INR > 1.5; PTT > 1.5) or those who are receiving anticoagulants.
  10. Thrombocytopenia (platelet count less than 100,000/mm3).
  11. Renal insufficiency (BUN > 30 mg/dlan/or serum creatinine > 1.9 mg/dl).
  12. Liver disease (bilirubin > 2.0 mg/dl and or > 2 fold increase of transaminases).
  13. Diagnosis of cancer made by lumpectomy or incisional biopsy.
  14. Contraindications to chemotherapy.
  15. Clinical tumor fixation to the pectoralis major muscle or presence of skin nodules, involvement of the nipple.
  16. Breast cancer with a high probability of extensive intra-ductal in situ disease (extensive DCIS or LCIS).
  17. Multicentric disease (no satellite tumors greater than 2 cm diameter and no greater than 1.5 cm from the primary tumor as measured from the edge of the satellite tumor to the nearest edge of the primary tumor).
  18. Prior history of collagen vascular disease.
  19. Previous participation in Celsion Corporation study 201 or 202.
  20. Subject has participated in an investigation drug or device trial 30 days prior to the screening visit or plans to enroll in an investigational drug or device trial at any time during this study. However current participation in another clinical study involving imaging is not exclusion.
  21. Subject has a history of drug or alcohol abuse in the last 12 months.
  22. Non-glandular breast cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2010-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Tumor Shrinkage (ultrasound) | Prior to Surgery, on average 4 months from the start of treatment
  Evaluate the efficiency of preoperative focused microwave thermotherapy as an adjunct to chemotherapy to increase the ultrasound-measured absolute mean tumor percent shrinkage by volume over that achieved by SOC preoperative chemotherapy.

SECONDARY OUTCOMES:
Conversion Rate to Breast Conservation (surgeon recommended) | Prior to Mastectomy Recommendation, on average 4 months from the start of treatment
  Evaluate the potential benefits of this combination treatment to increase the absolute rate for which the surgeon can recommend breast conservation (lumpectomy or partial mastectomy) over that achieved using standard of care preoperative chemotherapy alone.
Tumor Shrinkage (Clinical) | Prior to Surgery, on average 4 months from the start of treatment
  Evaluate the potential benefits of this combination treatment to increase the clinical (caliper-measured) absolute mean tumor shrinkage by area over that achieved by SOC preoperative chemotherapy
Tumor Shrinkage (Mammography) | Prior to Surgery, on average 4 months from the start of treatment
  Evaluate the potential benefits of the combination treatment to increase the absolute mean tumor shrinkage by area on mammography over the achieved by SOC preoperative chemotherapy
Tumor Shrinkage (MRI) | Prior to Surgery, on average 4 months from the start of treatment
  Evaluate the potential benefits of this combination treatment to increase the absolute mean tumor shrinkage by volume based on magnetic resonance imaging (MRI) over that achieved by SOC preoperative chemotherapy.
Tumor Necrosis (pathology) | After Surgery, on average 5 months from the start of treatment
  Evaluate the potential benefits of this combination treatment to increase the absolute mean percent localized pathologic tumor cell kill by volume over that achieved by SOC preoperative chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: William C. Dooley, MD, Principal Investigator — University of Oklahoma; John Keyserlingk, MD, Principal Investigator — Centre Medical Ville-Marie
Locations (2):
- Dr. William Dooley, Oklahoma City, Oklahoma, United States
- Ville-Marie Medical Centre, Montreal, Quebec, Canada

REFERENCES:
- [Background] Vargas HI; Dooley WC; Fenn AJ; Tomaselli MB; and Harness JK. Study of preoperative focused microwave phased array thermotherapy in combination with neoadjuvant anthracycline-based chemotherapy for large breast carcinomas. Cancer Therapy. 2007;5B:401-408. Available; http://www.cancer-therapy.org/CT5B/pdf/45._Vargas_et_al,_401-408.pdf. Accessed November 25, 2007. (background for protocol)
- [Background] Dooley WC, Vargas HI, Fenn AJ, Tomaselli MB, Harness JK. Focused microwave thermotherapy for preoperative treatment of invasive breast cancer: a review of clinical studies. Ann Surg Oncol. 2010 Apr;17(4):1076-93. doi: 10.1245/s10434-009-0872-z. Epub 2009 Dec 22. PMID 20033319